CLINICAL TRIAL: NCT05204134
Title: Adaptation of Insulin Delivery Settings to Improve Clinical Outcomes With AID Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-0009348
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; Control-IQ Technology; automated insulin dosing; automated insulin delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Control-IQ Technology with Algorithm Derived Initial Profile Settings and Regular Updates (Experimental): After CGM run-in, participants will begin use of Control-IQ technology with algorithm derived initial insulin delivery settings, then have regular settings updates from the algorithm through 13 weeks of use.
  Interventions: Device: Automated Insulin Delivery Settings Initialization and Adaptation Algorithm

INTERVENTIONS:
Device: Automated Insulin Delivery Settings Initialization and Adaptation Algorithm — All participants wearing the t:slim X2 insulin pump with Control-IQ technology, and wearing the Dexcom G6 sensor, will have algorithm derived insulin delivery profile settings initialization and updates at regular intervals.

SUMMARY:
Obtain preliminary safety and performance data on a settings initialization and adaptation algorithm used in conjunction with closed-loop control.

DETAILED DESCRIPTION:
This feasibility study is a prospective, single arm, single center study with a run-in phase, followed by 13 weeks of Control-IQ technology use. By using an algorithm to more accurately initialize insulin delivery settings and adapt them over time, faster than typical HCP visits, users onboarding from multiple daily injections (MDI) will reach optimal glycemic outcomes faster.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ≥ age 18 years
* Clinical diagnosis of type 1 diabetes for at least one year
* Using a basal/bolus regimen by injection (MDI therapy)
* Total daily dose ≥10 units/day
* Willing to use only aspart (novolog) or lispro (humalog) U-100 insulin with the study pump.
* A1c ≥ 7.5% and ≤ 11% at screening
* Not pregnant or planning a pregnancy during the time period of the study.
* Has current glucagon product to treat severe hypoglycemia (injectable or nasal) at home (will provide prescription if they do not have one)
* Willingness to follow study procedures and a signed informed consent form

Exclusion Criteria:

* Two or more episodes of severe hypoglycemia (needing assistance) in the past 6 months
* Two or more episodes of diabetic ketoacidosis in the past 6 months
* Inpatient psychiatric treatment in the past 6 months
* History of drug abuse (defined as any illicit drug use) or history of alcohol abuse prior to screening or unwillingness to agree to abstain from illicit drugs throughout the study
* Significant chronic kidney disease or hemodialysis
* Significant liver disease
* History of adrenal insufficiency
* Hypothyroidism or hyperthyroidism that is not appropriately treated
* Other chronic disease/condition determined by investigator to interfere with participation in the study
* Use of glucocorticoids, beta blockers or other medications determined by investigator to interfere with study
* Use of long-acting insulin, inhaled insulin (Afrezza), or use of any non-insulin glucose lowering agents (i.e. SGLT-2 inhibitor) other than Metformin with the study pump
* Subject is pregnant or lactating or intending to become pregnant before or during participation in this study
* Investigator judgement that subject would not be able to complete the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan E Pinsker, MD, Study Chair — Tandem Diabetes Care, Inc.
Locations (1):
- Barbara Davis Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shah VN, Akturk HK, Trahan A, Piquette N, Wheatcroft A, Schertz E, Carmello K, Mueller L, White K, Fu L, Sassan-Katchalski R, Messer LH, Habif S, Constantin A, Pinsker JE. Safety and Feasibility Evaluation of Automated User Profile Settings Initialization and Adaptation With Control-IQ Technology. J Diabetes Sci Technol. 2024 Nov;18(6):1281-1287. doi: 10.1177/19322968241229074. Epub 2024 Feb 7. PMID 38323362

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study performed at a single clinical site, Barbara Davis Center, from March to September 2022.
Groups:
- Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates: Participants will begin use of Control-IQ technology with algorithm derived initial insulin delivery settings, then have regular settings updates from the algorithm through 13 weeks of use
Period: Overall Study
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Started | 33
Completed Run-In | 33
Completed | 29
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Male and female participants ≥ 18 years of age with type 1 diabetes, who were multiple daily injection (MDI) users, who have a baseline hemoglobin A1c at screening between 7.5 to 11%.
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 25
  More than one race | 3
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 33
HbA1c at Enrollment [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] | 8.5 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Severe Hypoglycemic Events
Description: Number of Severe Hypoglycemic Events (with altered mental status)
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: number of events
Groups:
- Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates: All participants wearing the t:slim X2 insulin pump with Control-IQ technology, and wearing the Dexcom G6 sensor, will have algorithm derived insulin delivery profile settings initialization and updates at regular intervals over 13 weeks.
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
number of events
  MDI Run-In with CGM (2 Weeks) | 0 (0)
  Control-IQ with Adaptation (13 Weeks) | 0.06 (0.35)

2. Primary Outcome: Diabetic Ketoacidosis Events
Description: Number of Diabetic Ketoacidosis events as defined by the Diabetes Control and Complications Trial (DCCT)
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
number of events
  MDI Run-In with CGM (2 Weeks) | 0 (0)
  Control-IQ with Adaptation (13 Weeks) | 0 (0)

3. Secondary Outcome: Percent Time < 54 mg/dL, Overall
Description: CGM percent time < 54 mg/dL, Overall Study Participation
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
percentage of time
  MDI Run-In with CGM (2 Weeks) | 0.3 [0.1 to 0.7]
  Control-IQ with Adaptation (at 13 Weeks) | 0.2 [0.1 to 0.3]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p = 0.06, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Percent Time < 54 mg/dL, Daytime Outcomes
Description: CGM percent time < 54 mg/dL, Daytime Outcomes between 06:00-00:00
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
percentage of time
  MDI Run-In with CGM (2 Weeks) | 0.2 [0.1 to 0.5]
  Control-IQ with Adaptation (at 13 Weeks) | 0.2 [0.0 to 0.3]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p = 0.11, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Percent Time < 54 mg/dL, Overnight Outcomes
Description: CGM percent time < 54 mg/dL, Overnight Outcomes between 00:00-06:00
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
percentage of time
  MDI Run-In with CGM (2 Weeks) | 0.2 [0.0 to 0.9]
  Control-IQ with Adaptation (at 13 Weeks) | 0.2 [0.0 to 0.3]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Percent Time < 70 mg/dL, Overall
Description: CGM percent time < 70 mg/dL, Overall Study Participation
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
percentage of time
  MDI Run-In with CGM (2 Weeks) | 1.8 [1.1 to 3.8]
  Control-IQ with Adaptation (at 13 Weeks) | 1.0 [0.8 to 1.7]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Percent Time < 70 mg/dL, Daytime Outcomes
Description: CGM percent time < 70 mg/dL, Daytime Outcomes between 06:00-00:00
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
percentage of time
  MDI Run-In with CGM (2 Weeks) | 1.5 [0.7 to 3.0]
  Control-IQ with Adaptation (at 13 Weeks) | 1.1 [0.8 to 1.9]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p = 0.26, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Percent Time < 70 mg/dL, Overnight Outcomes
Description: CGM percent time < 70 mg/dL, Overnight Outcomes between 00:00-06:00
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
percentage of time
  MDI Run-In with CGM (2 Weeks) | 2.1 [0.9 to 4.6]
  Control-IQ with Adaptation (at 13 Weeks) | 1.0 [0.6 to 1.5]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p = 0.005, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Percent of Time 70-140 mg/dL, Overall
Description: CGM percent time 70-140 mg/dL, Overall Study Participation
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
percentage of time
  MDI Run-In with CGM (2 Weeks) | 26.0 [22.7 to 31.4]
  Control-IQ with Adaptation (at 13 Weeks) | 39.2 [36.3 to 48.7]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Percent of Time 70-140 mg/dL, Daytime Outcomes
Description: CGM percent time 70-140 mg/dL, Daytime Outcomes between 06:00-00:00
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
percentage of time
  MDI Run-In with CGM (2 Weeks) | 23.8 [19.7 to 29.8]
  Control-IQ with Adaptation (at 13 Weeks) | 39.0 [33.1 to 46.3]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Percent of Time 70-140 mg/dL, Overnight Outcomes
Description: CGM percent time 70-140 mg/dL, Overnight Outcomes between 00:00-06:00
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
percentage of time
  MDI Run-In with CGM (2 Weeks) | 29.4 [20.8 to 38.2]
  Control-IQ with Adaptation (at 13 Weeks) | 45.0 [36.6 to 61.6]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Percent of Time 70-180 mg/dL, Overall
Description: CGM percent time 70-180 mg/dL, Overall Study Participation
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
percentage of time
  MDI Run-In with CGM (2 Weeks) | 45.7 [40.5 to 56.7]
  Control-IQ with Adaptation (at 13 Weeks) | 69.1 [61.8 to 73.1]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Comparison between 2 week run-in and 13 weeks Control-IQ use with adaptation; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Percent of Time 70-180 mg/dL, Daytime Outcomes
Description: CGM percent time 70-180 mg/dL, Daytime Outcomes between 06:00-00:00
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
percentage of time
  MDI Run-In with CGM (2 Weeks) | 45.5 [36.8 to 54.3]
  Control-IQ with Adaptation (at 13 Weeks) | 65.4 [60.4 to 73.6]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Percent of Time 70-180 mg/dL, Overnight Outcomes
Description: CGM percent time 70-180 mg/dL, Overnight Outcomes between 00:00-06:00
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
percentage of time
  MDI Run-In with CGM (2 Weeks) | 53.5 [36.3 to 64.0]
  Control-IQ with Adaptation (at 13 Weeks) | 74.9 [64.8 to 82.9]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Percent Time > 180 mg/dL, Overall
Description: CGM percent time > 180 mg/dL, Overall Study Participation
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
percentage of time
  MDI Run-In with CGM (2 Weeks) | 51.9 [42.3 to 57.1]
  Control-IQ with Adaptation (at 13 Weeks) | 29.5 [26.2 to 37.4]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Percent Time > 180 mg/dL, Daytime Outcomes
Description: CGM percent time > 180 mg/dL, Daytime Outcomes between 06:00-00:00
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
percentage of time
  MDI Run-In with CGM (2 Weeks) | 52.5 [44.0 to 60.9]
  Control-IQ with Adaptation (at 13 Weeks) | 34.2 [24.2 to 38.9]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Percent Time > 180 mg/dL, Overnight Outcomes
Description: CGM percent time > 180 mg/dL, Overnight Outcomes between 00:00-06:00
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
percentage of time
  MDI Run-In with CGM (2 Weeks) | 38.7 [35.4 to 61.1]
  Control-IQ with Adaptation (at 13 Weeks) | 24.6 [13.2 to 34.1]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Percent Time > 250 mg/dL, Overall
Description: CGM percent time > 250 mg/dL, Overall Study Participation
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
percentage of time
  MDI Run-In with CGM (2 Weeks) | 21.8 [12.9 to 26.3]
  Control-IQ with Adaptation (at 13 Weeks) | 7.7 [6.1 to 11.4]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Percent Time > 250 mg/dL, Daytime Outcomes
Description: CGM percent time > 250 mg/dL, Daytime Outcomes between 06:00-00:00
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
percentage of time
  MDI Run-In with CGM (2 Weeks) | 19.6 [11.2 to 29.4]
  Control-IQ with Adaptation (at 13 Weeks) | 8.5 [6.3 to 11.5]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Percent Time > 250 mg/dL, Overnight Outcomes
Description: CGM percent time > 250 mg/dL, Overnight Outcomes between 00:00-06:00
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
percentage of time
  MDI Run-In with CGM (2 Weeks) | 20.1 [8.5 to 27.1]
  Control-IQ with Adaptation (at 13 Weeks) | 6.0 [3.7 to 10.6]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Median Sensor Glucose
Description: CGM-measured median glucose (mg/dL)
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
mg/dL
  MDI Run-In with CGM (2 Weeks) | 185.0 [165.0 to 196.0]
  Control-IQ with Adaptation (at 13 Weeks) | 149.0 [138.0 to 157.0]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Total Daily Insulin Use
Description: Total Daily Insulin Use (Units/Day)
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: units/day
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
units/day
  MDI Run-In with CGM (2 Weeks) | 55.0 [40.8 to 71.3]
  Control-IQ with Adaptation (at 13 Weeks) | 61.5 [40.4 to 79.9]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p = 0.17, Wilcoxon (Mann-Whitney)

23. Secondary Outcome: Total Daily Bolus Insulin Use
Description: Total Daily Bolus Insulin Use (units/day)
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: units/day
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
units/day
  MDI Run-In with CGM (2 Weeks) | 23.0 [19.0 to 25.0]
  Control-IQ with Adaptation (at 13 Weeks) | 25.3 [19.5 to 38.1]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney)

24. Secondary Outcome: Total Daily Basal Insulin Use
Description: Total Daily Basal Insulin Use (units/day)
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: units/day
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
units/day
  MDI Run-In with CGM (2 Weeks) | 32.5 [20.8 to 44.5]
  Control-IQ with Adaptation (at 13 Weeks) | 30.1 [17.2 to 44.9]
Statistical Analysis 1: Comparison: Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates; Test type: Superiority; p = 0.69, Wilcoxon (Mann-Whitney)

25. Secondary Outcome: Physician Overrides/Physician Initiated Changes in Pump Settings
Description: Number of physician overrides/physician initiated changes in pump settings during the entire study.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 33
number of events | 0.21 (0.42)

26. Secondary Outcome: Device Impact Score, as Reported on the Diabetes Impact and Satisfaction (DIDS) Scale at Study Completion
Description: The Diabetes Impact and Satisfaction (DIDS) scale is an 11-item questionnaire focused on satisfaction related to insulin delivery devices (e.g., trust and ease of use) and diabetes- elated impact on daily life, such as worry around hypoglycemia and sleep interruptions. The last 4 questions assess diabetes impact on a scale of 1-10 (1=Never, 10=always), with a lower score means a better outcome. Mean score for overall diabetes impact is reported after 13 weeks using the system with adaptive therapy settings
Time Frame: 13 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 29
units on a scale | 3.5 (2.2)

27. Secondary Outcome: Device Satisfaction Score, as Reported on the the Diabetes Impact and Satisfaction (DIDS) Scale at Study Completion
Description: The Diabetes Impact and Satisfaction (DIDS) scale is an 11-item questionnaire focused on satisfaction related to insulin delivery devices (e.g., trust and ease of use) and diabetes- elated impact on daily life, such as worry around hypoglycemia and sleep interruptions. The first 7 questions assess device satisfaction on a scale of 1-10 (1=strongly disagree, 10=strongly agree), with a higher score means a better outcome. Mean score for overall device satisfaction is reported after 13 weeks using the system with adaptive therapy settings
Time Frame: 13 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
Number analyzed (Participants) | 29
units on a scale | 8.9 (1.1)

ADVERSE EVENTS:
Time Frame: 15 weeks
Groups:
- MDI Run-In With CGM: Run-In with MDI therapy and CGM for 2 weeks.
- Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates: All participants wearing the t:slim X2 insulin pump with Control-IQ technology, and wearing the Dexcom G6 sensor, will have algorithm derived insulin delivery profile settings initialization and updates at regular intervals through 13 weeks of use.
Arm/Group | MDI Run-In With CGM | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 2/33
Other Adverse Events (participants affected / at risk) | 0/33 | 8/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MDI Run-In With CGM (N=33) | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates (N=33)
Severe Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (2) — The event required assistance of another person due to altered consciousness, and required another person to actively administer carbohydrate, glucagon, or other resuscitative actions.
Pancreatitis (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MDI Run-In With CGM (N=33) | Control-IQ Technology With Algorithm Derived Initial Profile Settings and Regular Updates (N=33)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Ketonemia (Endocrine disorders) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3)
Edema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT05204134/Prot_SAP_000.pdf